CLINICAL TRIAL: NCT03281291
Title: Molecular Detection and Genotyping of Plasmodium Falciparum Parasites in Young African Children After Immunization With RTS,S/AS01E Malaria Vaccine. An Ancillary Study Protocol to GlaxoSmithKline Phase IIb RTS,S/AS01E Malaria Vaccine Trial (Study Number 204889) Entitled, "Efficacy, Safety and Immunogenicity Study of GSK Biologicals' Candidate Malaria Vaccine (SB257049) Evaluating Schedules With or Without Fractional Doses, Early Dose 4 and Yearly Doses, in Children 5-17 Months of Age.
Brief Title: Study to Assess the Vaccine Efficacy Against Malaria Infection, in Children Immunized With the Primary and Yearly Booster of the RTS,S/AS01E Vaccine, as Part of Their Participation in the Malaria-094 (204889/NCT03276962) Study.
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 206213
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Malaria
Keywords: malaria vaccine; infants; malaria; RTS,S/AS01; falciparum; genomics; efficacy
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- R012-20 Group: Participants received a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2 and Month 20 of study NCT03276962.
- R012-14-mD Group: Participants received a full dose of RTS,S/AS01E at Month 0, Month 1, Month 2, Month 14, Month 26 and Month 38 of study NCT03276962.
- Fx012-14-mFxD Group: Participants received a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 2, Month 14, Month 26 and Month 38 of study NCT03276962.
- Fx017-mFxD Group: Participants received a full dose of RTS,S/AS01E at Month 0 and Month 1, and RTS,S/AS01E 1/5th dose at Month 7, Month 20 and Month 32 of study NCT03276962.
- Control Group: Participants received rabies vaccine at Month 0, Month 1 and Month 2 of study NCT03276962.

SUMMARY:
The aim of this study was to evaluate the effectiveness of the RTS,S/AS01E malaria vaccine against both clinical and asymptomatic malaria infections by detecting Plasmodium falciparum (P. falciparum) parasites in blood samples collected from children who received the primary and yearly booster doses of the RTS,S/AS01E vaccine, as part of their participation in the Malaria-094 parent clinical study. The genomic analysis was conducted on parasites found in blood spot samples from children aged 5-17 months, who were vaccinated according to different dosage and schedule regimens as part of the Malaria-094 parent clinical study.

DETAILED DESCRIPTION:
This genotyping study of malaria parasites, collected from serial blood samples following RTS,S/AS01E immunization, assessed vaccine efficacy using molecular genetic data. The study aimed to identify the first infections post-vaccination and distinguish new infections from existing ones through an amplicon sequencing-based strategy. This involved deep sequencing of small, highly variable regions of the parasite genome, enabling both: 1. Highly sensitive detection of parasitemia (similar to conventional polymerase chain reaction [PCR]-based detection), and 2. Identification of genetically distinct parasite populations within or between affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participants' parent(s)/LAR(s) who, in the opinion of the investigator, complied with the requirements of the protocol (e.g. return for follow-up visits).
* Signed or thumb-printed and witnessed informed consent obtained from the parent(s)/LAR(s) of the participant prior to performance of any study specific procedure. Where parent(s)/LAR(s) were illiterate, the consent form was countersigned by an independent witness.
* A male or female between, and including, five and 17 months of age at the time of the first vaccination.
* Healthy participants as established by medical history and clinical examination before entering into the study.
* Previously received three documented doses of diphtheria, tetanus, pertussis, hepatitis B vaccine (DTPHepB), and at least three doses of oral polio vaccine.

Exclusion Criteria:

* Child in care.
* Use of a drug or vaccine that is not approved for that indication (by one of the following regulatory authorities: Food and Drug Administration [FDA; USA] or European Union member state or WHO [with respect to prequalification]) other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -29 to Day 0), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would have made the intramuscular injection unsafe.

Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this meant prednisone (0.5 mg/kg/day (for pediatric participants) or equivalent. Inhaled and topical steroids are allowed.

* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting seven days before each dose and ending seven days after each dose of vaccine administration.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or was to be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* History of anaphylaxis post-vaccination.
* History of any, or documented, serious adverse reaction to rabies vaccination.
* Contraindication to rabies vaccination (Rabipur is contraindicated in participants with a history of a severe hypersensitivity to any of the ingredients in the vaccine. Note that the vaccine contains polygeline and residues of chicken proteins, and may contain traces of neomycin, chlortetracycline and amphotericin B).
* Major congenital defects.
* Serious chronic illness.
* Children with a past history of a neurological disorder or atypical febrile seizure (a febrile seizure is atypical if it meets one of the following criteria: not associated with fever; lasts > 5 minutes; focal (not generalized); followed by transient or persistent neurological abnormality; occurs in a child < 6 months of age).
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature ≥ 37.5°C/99.5°F for oral, axillary or tympanic route, or ≥ 38.0°C/100.4°F for rectal route.
* Participants with a minor illness (such as mild diarrhea, mild upper respiratory infection) without fever may have been enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products during the period starting three months before the first dose of study vaccine or planned administration during the study period.
* Moderate or severe malnutrition at screening defined as weight for age or weight for height Z-score < -2.
* Hemoglobin concentration < 8 g/dl at screening.
* Same sex twins (to avoid misidentification).
* Maternal death.
* Prior receipt of an investigational malaria vaccine.

Ages: 5 Months to 17 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2023-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Kumasi, Ghana
- GSK Investigational Site, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

REFERENCES:
- [Background] Juraska M, Early AM, Li L, Schaffner SF, Lievens M, Khorgade A, Simpkins B, Hejazi NS, Benkeser D, Wang Q, Mercer LD, Adjei S, Agbenyega T, Anderson S, Ansong D, Bii DK, Buabeng PBY, English S, Fitzgerald N, Grimsby J, Kariuki SK, Otieno K, Roman F, Samuels AM, Westercamp N, Ockenhouse CF, Ofori-Anyinam O, Lee CK, MacInnis BL, Wirth DF, Gilbert PB, Neafsey DE. Genotypic analysis of RTS,S/AS01E malaria vaccine efficacy against parasite infection as a function of dosage regimen and baseline malaria infection status in children aged 5-17 months in Ghana and Kenya: a longitudinal phase 2b randomised controlled trial. Lancet Infect Dis. 2024 Sep;24(9):1025-1036. doi: 10.1016/S1473-3099(24)00179-8. Epub 2024 May 6. PMID 38723650

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is an ancillary study of the Malaria-094 study (204889/NCT03276962). Consequently, the data reported in the Participant Flow and Baseline Characteristics sections were collected from participants from that study.
Pre-assignment Details: As pre-specified in the analysis plan, efficacy outcome measures corresponding to vaccine efficacy against first new infection (ATP Cohort) and vaccine efficacy against all new infections (ATP Cohort), presented data for the R012-20 + R012-14-mD Pooled Group because the interventional strategy (1st dose at Month 0, 2nd dose at Month 1, 3rd dose at Month 2) was the same for both the R012-20 Group and the R012-14-mD Group until Month 14.
Period: Overall Study
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Started | 298 | 294 | 304 | 311 | 293
Completed | 229 | 232 | 242 | 247 | 237
Not Completed | 69 | 62 | 62 | 64 | 56
Not completed — Serious Adverse Event And/Or pIMD | 2 | 1 | 0 | 4 | 1
Not completed — Protocol Deviation | 2 | 0 | 1 | 2 | 1
Not completed — Consent Withdrawal, Not Due To An Adverse Event/A Serious Adverse Event | 29 | 21 | 13 | 21 | 16
Not completed — Migrated / Moved From The Study Area | 26 | 28 | 44 | 29 | 27
Not completed — Lost to Follow-up | 10 | 10 | 4 | 6 | 10
Not completed — Other | 0 | 2 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Blood samples collected
Groups:
- Total: Total of all reporting groups
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group | Total
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293 | 1500
Number analyzed (Blood samples collected) | 8859 | 8761 | 9140 | 9392 | 9207 | 45359
Age, Continuous [Mean (Standard Deviation); unit: Months] | 10.2 (3.9) | 10.3 (3.8) | 10.5 (4.0) | 10.2 (3.8) | 10.5 (3.9) | 10.3 (3.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 155 | 172 | 163 | 152 | 761
  Male | 179 | 139 | 132 | 148 | 141 | 739
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 298 | 294 | 304 | 311 | 293 | 1500

OUTCOME MEASURES:

1. Primary Outcome: Time From First Vaccination to the Detection of the First New Malaria Infection Through to the Month 20 Study Visit
Description: The number of days from the time origin in each analysis to the visit date associated with the first molecular detection of a new malaria infection.
  A new molecularly confirmed malaria infection was defined by a detected new infection from genomic analysis of dried blood spot samples originating either from active monthly screening for infection or from unscheduled visits intended for the assessment of clinical malaria.
Time Frame: Up to 20 months post Dose 1
Population: The analysis was performed on the Total Vaccinated Cohort (TVC) which included all the participants who received at least one dose of study vaccine per Malaria-094 protocol.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Weeks | 43.1 [15.1 to 85.9] | 43.9 [17.4 to 86.4] | 39 [19.4 to 79.3] | 39 [15.7 to 87.7] | 31.9 [10.4 to 64.9]
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; Comparison of vaccine efficacy (VE) in the TVC against the first new genotypic infection, between enrollment and Month 20 visit, for R012-20 Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 29.7, 95% CI 2-sided [14.7 to 42.1] — VE = 1 minus the Hazard Ratio (HR). HR was defined as the ratio of relative risk of infection in the vaccinated group compared to the control group
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 20 visit, for R012-14-mD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 31.2, 95% CI 2-sided [16.4 to 43.3] — VE = 1 minus HR. HR was defined as the ratio of relative risk of infection in the vaccinated group compared to the control group
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 20 visit, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 24.6, 95% CI 2-sided [9.0 to 37.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 20 visit, for Fx017-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 28.8, 95% CI 2-sided [13.9 to 41.1] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Time From First Vaccination to the Detection of the First New Malaria Infection From 14 Days Post-Dose 3 Through to 12 Months Post-Dose 3
Description: as for outcome 1
Time Frame: From Month 2.5 to Month 14 for the R012-20 + R012-14-mD Pooled Group, the Fx012-14-mFxD Group and the Control Group, and from Month 7.5 to Month 19 for the Fx017-mFxD Group
Population: The analysis was performed on the According-To-Protocol (ATP) cohort, including participants who received the first three vaccinations per Malaria-094 protocol and were at risk for a molecularly confirmed infection 14 days after Dose 3. As pre-specified in the analysis plan, this outcome measure was reported for the R012-20 + R012-14-mD Pooled Group because both the R012-20 Group and R012-14-mD Group followed the same interventional strategy until Month 14.
Measure: Median (Inter-Quartile Range); unit: Weeks
Groups:
- R012-20 + R012-14-mD Pooled Group: Participants received full doses of RTS,S/AS01E at Month 0, Month 1, Month 2 and a full dose at Month 14, Month 20, Month 26 and Month 38 of study NCT03276962.
Arm/Group | R012-20 + R012-14-mD Pooled Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 523 | 271 | 273 | 265
Weeks | 40.6 [20.4 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 36.7 [21.9 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 38.6 [12.6 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 28.7 [10.6 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring.
Statistical Analysis 1: Comparison: R012-20 + R012-14-mD Pooled Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 2.5 and 14, for R012-20 + R012-14-mD Pooled Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 42.8, 95% CI 2-sided [30.7 to 52.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Fx012-14-mFxD Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 2.5 and 14, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 36.7, 95% CI 2-sided [21.2 to 49.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Fx017-mFxD Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 7.5 and 19, for Fx017-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 41.4, 95% CI 2-sided [26.7 to 53.1] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Time From First Vaccination to the Detection of the First New Malaria Infection Through to the Month 32 Study Visit
Description: as for outcome 1
Time Frame: Up to 32 months post Dose 1
Population: The analysis was performed on the TVC which included all the participants who received at least one dose of study vaccine per Malaria-094 protocol.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Weeks | 42.4 [12.6 to 97.1] | 42.7 [12.7 to 97.7] | 38.9 [19.6 to 79.3] | 37.7 [14.7 to 94] | 31 [10.3 to 64]
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 32 visit, for R012-20 Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 29.6, 95% CI 2-sided [15.4 to 41.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 32 visit, for R012-14-mD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 30.6, 95% CI 2-sided [16.6 to 42.2] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 32 visit, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 27.4, 95% CI 2-sided [13.1 to 39.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; Comparison of vaccine efficacy in the TVC against the first new genotypic infection, between enrollment and Month 32 visit, for Fx017-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 26.3, 95% CI 2-sided [11.9 to 38.3] — [estimate comment as in outcome 1, analysis 2]

4. Primary Outcome: Time From First Vaccination to the Detection of the First New Malaria Infection From 14 Days Post-Dose 3 Through to 24 Months Post-Dose 3
Description: as for outcome 1
Time Frame: From Month 2.5 to Month 26 for the R012-20 Group, the R012-14-mD Group, the Fx012-14-mFxD Group and the Control Group, and from Month 7.5 to Month 31 for the Fx017-mFxD Group
Population: The analysis was performed on the ATP cohort which included all participants who received the first three vaccinations according to the Malaria-094 protocol procedures and who were observed to be at risk for a molecularly confirmed malaria infection at 14 days post-Dose 3.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 259 | 264 | 271 | 273 | 265
Weeks | 40.3 [20 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 42 [20.3 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 36.7 [21.9 to 83.7] | 38.4 [12.6 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring. | 28.7 [10.4 to NA] — The upper limit represents the time at which 75% of the population has experienced the event. This was not reached because, by the end of the study, less than 75% of the participants have experienced the event, therefore, this value could not be estimated. Q3 values are missing due to Kaplan Meier estimates accounting for right censoring.
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 2.5 and 26, for R012-20 Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 41.8, 95% CI 2-sided [28.6 to 52.5] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 2.5 and 26, for R012-14-mD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 39.9, 95% CI 2-sided [26.8 to 50.6] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 2.5 and 26, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 33.6, 95% CI 2-sided [19.3 to 45.3] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; Comparison of vaccine efficacy in the ATP cohort against the first new genotypic infection, between months 7.5 and 31, for Fx017-mFxD Group vs Control Group; Test type: Other; Regression, Cox; Vaccine Efficacy = 40.6, 95% CI 2-sided [27.2 to 51.5] — [estimate comment as in outcome 1, analysis 2]

5. Primary Outcome: Number of Molecularly Confirmed New Malaria Infections Through to the Month 20 Study Visit
Description: A new molecularly confirmed malaria infection was defined by a detected new infection from genomic analysis of dried blood spot samples originating either from active monthly screening for infection or from unscheduled visits intended for the assessment of clinical malaria.
Time Frame: Up to 20 months post Dose 1
Population: as for outcome 3
Measure: Number; unit: Infections
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Infections | 758 | 558 | 605 | 673 | 996
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 20 visit, for R012-20 Group vs Control Group; Test type: Other; Wald Test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.500, 95% CI 2-sided [-1.979 to -1.022] — Additive difference was defined as the difference in the mean number of new molecularly confirmed malaria infections between each vaccine arm and the control arm
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 20 visit, for R012-14-mD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.544, 95% CI 2-sided [-2.027 to -1.061] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 20 visit, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.575, 95% CI 2-sided [-2.065 to -1.085] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 20 visit, for Fx017-mFxD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.110, 95% CI 2-sided [-1.635 to -0.586] — [estimate comment as in outcome 5, analysis 1]

6. Primary Outcome: Number of Molecularly Confirmed New Malaria Infections From 14 Days Post-Dose 3 Through to 12 Months Post-Dose 3
Description: as for outcome 5
Time Frame: as for outcome 2
Population: The analysis was performed on the ATP cohort which included all participants who received the first 3 vaccinations according to the Malaria-094 protocol and who were observed to be at risk for a molecularly confirmed malaria infection at 14 days post-Dose 3. As pre-specified in the analysis plan, this outcome measure was reported for the R012-20 + R012-14-mD Pooled Group because both the R012-20 Group and R012-14-mD Group followed the same interventional strategy until Month 14.
Measure: Number; unit: Infections
Arm/Group | R012-20 + R012-14-mD Pooled Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 523 | 271 | 273 | 265
Infections | 1825 | 337 | 368 | 477
Statistical Analysis 1: Comparison: R012-20 + R012-14-mD Pooled Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 2.5 to 14, for R012-20 + R012-14-mD Pooled Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -0.769, 95% CI 2-sided [-1.068 to -0.469] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: Fx012-14-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 2.5 to 14, for Fx012-14-mFxD groups vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -0.786, 95% CI 2-sided [-1.133 to -0.439] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fx017-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 7.5 to 19, for Fx017-mFxD groups vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.275, 95% CI 2-sided [-1.592 to -0.959] — [estimate comment as in outcome 5, analysis 1]

7. Primary Outcome: Number of Molecularly Confirmed New Malaria Infections Through to the Month 32 Study Visit
Description: as for outcome 5
Time Frame: Up to 32 months post Dose 1
Population: as for outcome 3
Measure: Number; unit: Infections
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 298 | 294 | 304 | 311 | 293
Infections | 1105 | 940 | 910 | 1029 | 1420
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 32 visit, for R012-20 Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -2.686, 95% CI 2-sided [-3.448 to -1.924] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 32 visit, for R012-14-mD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -2.452, 95% CI 2-sided [-3.217 to -1.686] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 32 visit, for Fx012-14-mFxD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -2.585, 95% CI 2-sided [-3.345 to -1.824] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the TVC between enrollment and Month 32 visit, for Fx017-mFxD Group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.897, 95% CI 2-sided [-2.726 to -1.067] — [estimate comment as in outcome 5, analysis 1]

8. Primary Outcome: Number of Molecularly Confirmed New Malaria Infections From 14 Days Post-Dose 3 Through to 24 Months Post-Dose 3
Description: as for outcome 5
Time Frame: as for outcome 4
Population: The analysis was performed on the ATP cohort which included all participants who received the first three vaccinations according to the Malaria-094 protocol procedures and who are observed to be at risk for a molecularly confirmed malaria infection at 14 days post-Dose 3.
Measure: Number; unit: Infections
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
Number analyzed (Participants) | 259 | 264 | 271 | 273 | 265
Infections | 804 | 728 | 704 | 836 | 1071
Statistical Analysis 1: Comparison: R012-20 Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 2.5 to 26, for R012-20 group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.633, 95% CI 2-sided [-2.252 to -1.015] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: R012-14-mD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 2.5 to 26, for R012-14 group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.997, 95% CI 2-sided [-2.601 to -1.393] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: Fx012-14-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 2.5 to 26, for Fx012-14-mFxD group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.776, 95% CI 2-sided [-2.399 to -1.153] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Fx017-mFxD Group vs Control Group; To detect a significant difference in the mean number of new molecularly confirmed malaria infections in the ATP cohort between months 7.5 to 31, for Fx017-mFxD group vs Control Group; Test type: Other; Wald test; Wald tests were used to test for additive differences in VE differing from zero and to obtain a 95% confidence interval; Additive difference = -1.843, 95% CI 2-sided [-2.527 to -1.158] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious Adverse Events, and Other Adverse Events were not monitored/assessed.
Description: As pre-specified in the protocol, the adverse events were collected under the Malaria-094 (204889/NCT03276962) study. Therefore, no safety assessment was conducted for the Malaria-095 (206213/NCT03281291) study. Since no safety data was assessed, the total number of participants at risk and affected by All-Cause Mortality, Serious Adverse Events, and Other Adverse Events is zero.
Arm/Group | R012-20 Group | R012-14-mD Group | Fx012-14-mFxD Group | Fx017-mFxD Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03281291/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT03281291/SAP_001.pdf